CLINICAL TRIAL: NCT06700629
Title: Preoperative Predictors of Distal Hypospadias Repair Outcome
Brief Title: Distal Hypospadias Repair Outcome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armia Ezzat Thabet Azer (Other)
Responsible Party: Sponsor-Investigator, Armia Ezzat Thabet Azer, Resident physician, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DPH repair outcome
Record Dates: First submitted 2024-09-10; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Distal Penile Hypospadias (Disorder)
Keywords: Penile Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DPH repair outcome (Other): Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): A. Preoperative preparation: All patients will be subjected to evaluation including: 1. Measurement of penile length and width (in cm). 2. The shape of glans. (clefted , incomplete ceft, flat) 3. Glans size is measured by cubic centimetres. 4. Presence or absence of chordee and its degree. 5. Urethral plate condition and it's length, width and surface area. 6. Condition of skin over the urethra. 7. Presence of penile torsion. All patients should undergo preoperative surgical fitness including; complete blood picture, prothrombin time, concentration and INR, ECG and renal function test. Prophylactic systemic antibiotics are given intraoperatively.
  Interventions: Procedure: Distal Penile Hypospadias (Disorder)

INTERVENTIONS:
Procedure: Distal Penile Hypospadias (Disorder) — Three operations which are Tubularized incised plate urethroplasty (TIP), Mathieu and meatal advancement and glanuplasty (MAGPI).
  A three experienced operators with number of operations done by each one more than one hundred operation in the last year.
  The operators will be fixed for each surgical technique as follows:
  1. Doctor (A) for Matheiu. ( 35 operations)
  2. Doctor (M) for MAGPI. ( 35 operations)
  3. Doctor (S) for TIP ( 35 operations). Tubularized incised plate urethroplasty:(3,6) Indication: for distal penile hypospadias with or without penile curvature with any width of the uretheral plate and also for any type of distal hypospadias associated with curvature.
  Key steps for this operation are as follows:
  Glans retraction using stay suture 4-0 or 5-0 silk. Uretheral catheter pass through hypospadic meatus to bladder. Parallel longitudenal incision is done 1-2mm proximal to hypospadic meatus. A circumferential incision is made 2-3 mm below coronal sulcus dorsally
  Other Names: Distal Penile Hypospadias repair outcome

SUMMARY:
Aim is : To define the preoperative parameters that may influence the results of distal hypospadias repair

DETAILED DESCRIPTION:
Hypospadias is a congenital deformity where the opening of the urethra (the meatus) is sited on the underside (ventral) part of the penis, anywhere from the glans to the perineum.

It occurs in 1 in 250 live male births. it is often associated with "hooded" foreskin and chordee (ventral curvature of the penis shaft).

Hypospadias can be classified according to the anatomical location of meatus:

Distal-anterior hypospadias (located on the glans or distal shaft of the penis and the most common type of hypospadias) Intermediate-middle (penile). Proximal-posterior (penoscrotal, scrotal, perineal).

Diagnosis includes a description of the local findings:

Position, shape and width of the orifice Presence of atretic urethra and division of corpus spongiosum Appearance of the preputial hood and scrotum Size of the penis Curvature of the penis on erection. Aim of hypospadias surgery :(2) Is to correct penile curvature,to form neo-urethera of an adequate size, to bring the neomeatus to the tip of glans, and offer satisfactory cosmetic results.

The ideal age at surgery for primary hypospadias repair is usually 6-18 months. The complication rate is about 10% in distal hypospadias repair.

Complications include:

1. uretherocutaneous fistula.
2. meatal stenosis.
3. urethral stricture.
4. Urethral diverticulum. After hypospadias repairs, long-term follow-up is necessary, up to adolescence, to detect urethral stricture, voiding dysfunction and recurrent penile curvature.

ELIGIBILITY:
Inclusion Criteria:

* Child with distal hypospadias, uncircumcised , without meatal stenosis and no previous surgery for hypospadias

Exclusion Criteria:

* Any surgical manipulation includes circumcision or meatotomy. Patient refusal to be enrolled in the research. Patient lost follow up in the first six months

Min Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of Distal Penile Hypospadias Repair | Six months postoperatively
  Functional Outcome of Distal Hypospadias Repair. Outcome Measure Title: Post-void Residual Volume (PVR) Measured via Abdominal Ultrasound Description: Assessment of urinary function through post-void residual volume using ultrasound, reported in milliliters (mL).
  Time Frame: six months postoperatively.

SECONDARY OUTCOMES:
Cosmetic outcome of Distal Penile Hypospadias Repair | Six months postoperatively
  Cosmetic Outcome of Distal Hypospadias Repair. Outcome Measure Title: Aesthetic Evaluation Based on Photographic Documentation Description: Assessment of cosmetic outcomes using photographs taken on postoperative days 0 (immediately after surgery), 3, and 5-7 (during catheter removal), scored on a 5-point Likert scale (1 = poor, 5 = excellent).
  Time Frame: Six months postoperatively.
Complication Rate Following Distal Hypospadias Repair | Weekly assessments during the first month and monthly assessments for the following five months postoperatively.
  Complication Rate Following Distal Hypospadias Repair. Outcome Measure Title: Frequency of Postoperative Complications
  Description: Detection and quantification of specific complications, including:
  Edema of the glans or penile skin. Hematoma. Infection. Wound dehiscence. Urethrocutaneous fistula. Meatal stenosis. Urethral stricture. Urethral diverticula. Data will be reported as the number and percentage of patients experiencing each complication.
  Time Frame: Weekly assessments during the first month and monthly assessments for the following five months postoperatively.
Patient-Reported Outcomes | Six months postoperatively
  Patient-Reported Outcomes. Outcome Measure Title: Satisfaction Score as Reported by Patients or Caregivers Description: Patients or their relatives will report satisfaction with surgical outcomes on a Visual Analog Scale (VAS) ranging from 0 (not satisfied) to 10 (very satisfied).
  Time Frame: Six months postoperatively.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty Of Medicine Assiut University, Asyut, Asyut Governorate
  - Noha Elabody, Asyut

REFERENCES:
- [Background] 1) Belman AB. Hypospadias and chordee. In: Belman AB, King LR, Kramer SA, eds. Clinical Pediatric Urology. 4th edn. London, Martin Dunitz, 2002, pp. 1061-1092. 2) Mouriquand OD, Mure PY. Hypospadias. In: Gearhart J, Rink R, Mouriquand PDE, eds. Pediatric Urology, Philadelphia, WB Saunders, 2001, pp. 713-728. 3) Snodgrass W (1994) Tubularized, incised plate urethroplasty for distal hypospadias 151: 464-465. 4) Duckett JW Jr, Kaplan GW, Woodard JR, Devine CJ Jr (1980) Panel: complications of hypospadias repair 7: 443-454. 5) Braga LHP, Lorenzo AJ, Pippi Salle JL. Tubularized incised plate urethroplasty for distal hypospadias: A literature review. Indian J Urol 2008 Apr; 24(2)219-25. 6) Allen TD,Spence HM: The Surgical Treatment Of Coronal hypospadias and related problems , J. Urol 100:504, 1968. 7) Holland AJA, Smith GHH, Ross Fl, et al. HOSE: an objective scoring system for evaluating the results of hypospadias surgery. BJU Int 2001;88:255-8. 8) Hinman F. Penis: Plastic operation. In: Atlas of urologic surgery 2nd ed. Philadelphia; WB Saunders, 1998:96-157. 9) Abdul-Ghafoor B, Al-Dabbagh H. Primary distal hypospadias repair: tubularized incised plate urethroplasty (Snodgrass) versus the perimeatal based flap (Mathieu). Iraqi J Com Med 2009; 23-1. Rabnowitz R. and Hulbert W.C: Meatal-based flap Mathieu procedure. Adult and Pediatric. Saunders, Philadelphia, pp 39-43, 1999